CLINICAL TRIAL: NCT00031655
Title: Nonmyeloablative Allogeneic Hematopoietic Cell Transplantation From HLA Matched Unrelated Donors for Treatment of Patients With High Risk Acute Lymphocytic Leukemia in Complete Remission - A Multicenter Trial
Brief Title: Reduced Intensity Donor Stem Cell Transplant in Treating Patients With High Risk Acute Lymphocytic Leukemia in Complete Remission
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Georges, George, Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Organization: Fred Hutchinson Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1623.00; NCI-2012-00580 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); P01CA018029 (NIH)
Record Dates: First submitted 2002-03-08; First posted 2003-01-27 (Estimated); Last update posted 2012-12-07 (Estimated); Status verified 2012-12

CONDITIONS: Adult Acute Lymphoblastic Leukemia in Remission; Childhood Acute Lymphoblastic Leukemia in Remission; Recurrent Adult Acute Lymphoblastic Leukemia; Recurrent Childhood Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Cyclosporine; Whole-Body Irradiation; fludarabine phosphate; Mycophenolic Acid; Peripheral Blood Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (nonmyeloablative allogeneic PBSCT) (Experimental): NONMYELOALATIVE CONDITIONING REGIMEN: Patients receive fludarabine phosphate IV on days -4 to -2 and undergo TBI on day 0.
  TRANSPLANTATION: Patients undergo allogeneic PBSCT on day 0. Patients with minimal residual disease may receive donor lymphocyte infusion IV.
  IMMUNOSUPPRESSION: Patients receive cyclosporine PO every 12 hours on days -3 to 100 with taper to day 177 and mycophenolate mofetil PO very 8 hours on days 0 to 40 with taper to day 96.
  Interventions: Procedure: nonmyeloablative allogeneic hematopoietic stem cell transplantation; Biological: donor lymphocytes; Drug: cyclosporine; Radiation: total-body irradiation; Drug: fludarabine phosphate; Drug: mycophenolate mofetil; Other: laboratory biomarker analysis; Procedure: peripheral blood stem cell transplantation

INTERVENTIONS:
Procedure: nonmyeloablative allogeneic hematopoietic stem cell transplantation — Undergo nonmyeloablative allogeneic PBSCT
Biological: donor lymphocytes — Given IV
Drug: cyclosporine — Given PO
  Other Names: ciclosporin; cyclosporin; cyclosporin A; CYSP; Sandimmune
Radiation: total-body irradiation — Undergo TBI
  Other Names: TBI
Drug: fludarabine phosphate — Given IV
  Other Names: 2-F-ara-AMP; Beneflur; Fludara
Drug: mycophenolate mofetil — Given PO
  Other Names: Cellcept; MMF
Other: laboratory biomarker analysis — Correlative studies
Procedure: peripheral blood stem cell transplantation — Undergo nonmyeloablative allogeneic PBSCT
  Other Names: PBPC transplantation; PBSC transplantation; peripheral blood progenitor cell transplantation; transplantation, peripheral blood stem cell

SUMMARY:
The reason for doing this study is to determine whether a new method of blood stem cell transplant (also known as bone marrow transplant) is able to treat acute lymphocytic leukemia. Blood stem cells are the "seed cells" necessary to make all blood cells. This new method of transplant uses a combination of low dose radiation and chemotherapy that may be less toxic and cause less harm than a conventional transplant. This lower dose transplant is called a "nonmyeloablative transplant". Researchers want to see if using less radiation and less chemotherapy combined with new immune suppressing drugs after the transplant will help a stem cell transplant to work. Researchers hope that this treatment will cure acute lymphocytic leukemia with fewer side effects. Researchers are hoping to see a mixture of recipient and donor blood cells after transplant. This mixture of donor and recipient blood cells is called "mixed chimerism". Researchers hope that donor cells will attack and eliminate the leukemia. This is called the "graft-versus-leukemia" effect. In addition, after the transplant, white blood cells from the donor may be given to enhance or "boost" the graft-versus-leukemia effect, and hopefully remove all remaining cancer cells. This study is being done because at the present time blood stem cell transplantation (or bone marrow transplantation) is the only known curative therapy for acute lymphocytic leukemia. Because of age or underlying health status acute lymphocytic leukemia patients have a higher likelihood of experiencing severe harm from a conventional blood stem cell transplant. Researchers are doing this study to see if this new nonmyeloablative method of low dose radiation and low dose chemotherapy given before transplant and immune suppressive drugs after transplant will help make the transplant safer and also cure acute lymphocytic leukemia

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine if a one-year disease-free survival (DFS) of > 25% can be achieved among adult patients with high risk acute lymphocytic leukemia (ALL) in complete remission (CR) who undergo nonmyeloablative allografting.

II. To determine if a one-year DFS of >= 40% can be achieved among pediatric patients with high risk ALL in CR who undergo nonmyeloablative allografting.

SECONDARY OBJECTIVES:

I. To determine if a day +200 transplant-related mortality (TRM) of < 25% can be achieved among patients with high risk ALL in CR who undergo nonmyeloablative allografting.

II. To evaluate the efficacy and toxicity of donor lymphocyte infusion (DLI) in the treatment of minimal residue disease (MRD) after nonmyeloablative allografting for patients with high risk ALL in CR.

OUTLINE:

NONMYELOALATIVE CONDITIONING REGIMEN: Patients receive fludarabine phosphate intravenously (IV) on days -4 to -2 and undergo total body irradiation (TBI) on day 0.

TRANSPLANTATION: Patients undergo allogeneic peripheral blood stem cell transplantation (PBSCT) on day 0. Patients with minimal residual disease may receive donor lymphocyte infusion IV.

IMMUNOSUPPRESSION: Patients receive cyclosporine orally (PO) every 12 hours on days -3 to 100 with taper to day 177 and mycophenolate mofetil PO very 8 hours on days 0 to 40 with taper to day 96.

After completion of study treatment, patients are followed up at days 28, 56, 84, 120, 180, and 360; at 18 months; and annually for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* ADULT PATIENTS:
* Patients 50-75 years old with high risk ALL in first CR (CR1) or ALL in CR >= second CR (CR2)
* Patients >= 18 years old and < 50 years old with high risk ALL in CR1 who are not eligible for a conventional allogeneic transplantation based on general medical condition
* Patients >= 18 years old and < 50 years old with high risk ALL in CR1 who refuse a conventional allogeneic transplant
* Patients >= 18 years old and < 50 years old with ALL in CR >= CR2 who are not eligible for a conventional allogeneic transplantation based on general medical condition
* Patients >= 18 years old and < 50 years old with high risk ALL in CR >= CR2 who refuse a conventional allogeneic transplant
* CR is defined as < 5% blasts by morphology on a bone marrow aspirate and the absence of peripheral blasts
* High risk adult ALL in CR1 includes those patients with one or more of the following:

  * Age >=30 years
  * Non T-cell phenotype
  * Cytogenetic abnormalities including t(9;22), t(4;11), trisomy 8, or monosomy 7
  * Failure to achieve CR after 4 weeks of induction chemotherapy
* PEDIATRIC PATIENTS:
* Patients < 18 years old with ALL in high risk CR1 who are not candidates for conventional allogeneic transplantation based on general medical condition
* Patients < 18 years old with ALL in CR >= CR2 who are not candidates for conventional allogeneic transplantation based on general medical condition
* Patients < 12 years old require approval by the Fred Hutchinson Cancer Research Center (FHCRC) principal investigator prior to enrollment
* CR is defined as < 5% blasts by morphology on a bone marrow aspirate and absence of peripheral blasts
* High risk pediatric ALL in CR1 includes those patients with one or more of the following:

  * Cytogenetic abnormalities including:

    * t(9;22) with a white blood cell (WBC) >= 25,000 at diagnosis or
    * t(4;11) in patients < 1 year old and >= 10 years old or
    * Hypodiploidy (< 45 chromosomes)
  * Failure to achieve CR after 4 weeks of induction chemotherapy
  * Persistent peripheral blasts after one week of induction chemotherapy
* DONOR: FHCRC matching Grade 2.1: Unrelated donors who are prospectively:

  * Matched for human leukocyte antigen (HLA)-DRB1 and DQB1 alleles (must be defined by high resolution typing) and
  * Only a single allele disparity will be allowed for HLA-A, B, or C as defined by high resolution typing
* DONOR: A positive anti-donor cytotoxic crossmatch is an absolute donor exclusion; donors are excluded when preexisting immunoreactivity is identified that would jeopardize donor hematopoietic cell engraftment; this determination is based on the standard practice of the individual institution; the recommended procedure for patients with 10 of 10 HLA allele level (phenotypic) match is to obtain a panel reactive antibody (PRA) screens to class I and class II antigens for all patients before hematopoietic cell transplantation (HCT); if the PRA shows > 10% activity, then flow cytometric or B and T cell cytotoxic cross matches should be obtained; the donor should be excluded if any of the cytotoxic cross match assays are positive; for those patients with an HLA class I allele mismatch, flow cytometric or B and T cell cytotoxic cross matches should be obtained regardless of the PRA results
* DONOR: Patient and donor pairs homozygous at a mismatched allele are considered a two-allele mismatch, i.e., the patient is A*0101 and the donor is A*0102, and this type of mismatch is not allowed
* DONOR: Donor must consent to peripheral blood stem cell (PBSC) mobilization with filgrastim (G-CSF) arranged through the National Marrow Donor Program (NMDP) or other donor centers

Exclusion Criteria:

* Active central nervous system (CNS) disease
* Presence of circulating leukemic blasts (in the peripheral blood) detected by standard pathology
* Fertile men or women unwilling to use contraceptive techniques during and for 12 months following treatment
* Pregnancy or breastfeeding
* Human immunodeficiency virus (HIV) seropositivity
* ORGAN DYSFUNCTION, ADULT CRITERIA:
* Requiring supplementary continuous oxygen OR diffusing capacity of the lung for carbon monoxide (DLCO) < 40%
* Cardiac ejection fraction < 35%
* Patients with clinical or laboratory evidence of liver disease would be evaluated for the cause of liver disease, its clinical severity in terms of liver function, and the degree of portal hypertension; patients will be excluded if they are found to have fulminant liver failure, cirrhosis of the liver with evidence of portal hypertension, alcoholic hepatitis, esophageal varices, a history of bleeding esophageal varices, hepatic encephalopathy, uncorrectable hepatic synthetic dysfunction evinced by prolongation of the prothrombin time, ascites related to portal hypertension, bridging fibrosis, bacterial or fungal liver abscess, biliary obstruction, chronic viral hepatitis with total serum bilirubin > 3 mg/dL, and symptomatic biliary disease
* Karnofsky performance score < 50
* ORGAN DYSFUNCTION, PEDIATRIC CRITERIA:
* Lansky play-performance score < 40
* Patients with active non-hematologic malignancies (except non-melanoma skin cancers)
* Patients with a history of non-hematologic malignancies (except non-melanoma skin cancers) currently in a complete remission, who are less than 5 years from the time of complete remission, and have a > 20% risk of disease recurrence

Max Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2001-09; Primary Completion 2006-08 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Leukemia-free survival | 1 year
  Incidence of survival without relapse. Kaplan-Meier estimates will be used to estimate one-year leukemia-free survival.

SECONDARY OUTCOMES:
Transplant-related mortality | Day +200
Transplant-related mortality | 1 year
Efficacy of DLI for the elimination of MRD | Up to day 120
Toxicity of DLT, graded using a modified version of the National Cancer Institute (NCI) Common Toxicity Criteria | Up to 5 years
Overall survival | 1 year
Incidence of relapse | 1 year
Incidence of rejection | 1 year
Incidence of acute grade II-IV graft-versus-host disease (GVHD) and chronic GVHD, graded using a modified version of the National Cancer Institute (NCI) Common Toxicity Criteria | Up to 5 years
Karnofsky performance score and Lansky performance score | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: George Georges, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (3):
- United States (3):
  - Oregon Health and Sciences University, Portland, Oregon
  - Veterans Affairs Puget Sound Healthcare System, Seattle, Washington
  - Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington

REFERENCES:
- [Derived] Cooper JP, Storer BE, Granot N, Gyurkocza B, Sorror ML, Chauncey TR, Shizuru J, Franke GN, Maris MB, Boyer M, Bruno B, Sahebi F, Langston AA, Hari P, Agura ED, Lykke Petersen S, Maziarz RT, Bethge W, Asch J, Gutman JA, Olesen G, Yeager AM, Hubel K, Hogan WJ, Maloney DG, Mielcarek M, Martin PJ, Flowers MED, Georges GE, Woolfrey AE, Deeg JH, Scott BL, McDonald GB, Storb R, Sandmaier BM. Allogeneic hematopoietic cell transplantation with non-myeloablative conditioning for patients with hematologic malignancies: Improved outcomes over two decades. Haematologica. 2021 Jun 1;106(6):1599-1607. doi: 10.3324/haematol.2020.248187. PMID 32499241